CLINICAL TRIAL: NCT05801133
Title: Pifenidone is Used to Reduce Radiation Lung Injury in Lung Cancer Patients Previously Treated With Immune Checkpoint Inhibitors: A Single-arm, Open-label, Phase II Study
Brief Title: Pifenidone Prophylactic Therapy for Radiation Lung Injury in Patients Who Have Previously Received Immune Checkpoint Inhibitors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, professor, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBRT-2023-01
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pirfenidone combined with radiotherapy (Experimental): Pirfenidone: synchronized with RT, 200 mg TID in the first week, 300 mg TID in the second week, and maintenance treatment of 400 mg TID from the third week until 3 months
  Radiotherapy: no limitation, TD≥50Gy (BED/ α/β： 10）
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — 200 mg TID in the first week, 300 mg TID in the second week, and maintenance treatment of 400 mg TID from the third week until 3 months
  Other Names: PFD; AiSiRui

SUMMARY:
Patients with advanced lung cancer who have previously received immunocheckpoint inhibitor therapy, undergone chest radiation therapy again have developed radiation induced lung injury. Pirfenidone has anti-inflammatory and anti fibrosis effects. This study is intended to evaluate the effectiveness of pirfenidone combined with radiotherapy in the prevention of radiation pneumonitis.

ELIGIBILITY:
Inclusion Criteria:

1. The patients joined the study voluntarily and signed an informed consent form (ICF). They had good compliance and cooperated with follow-up;
2. Patients with lung cancer who had received at least 2 cycles of immunomonotherapy or combination systemic therapy (including PD-1 or PD-L1 immunocheckpoint inhibitors) within 6 months;
3. Age ≥ 18 years, no gender limit;
4. ECOG PS score: 0～1;
5. The expected survival time ≥ 3 months;
6. Use appropriate methods of contraception or surgical sterilization during treatment and for 3 years after treatment for men and women of reproductive age；
7. Appropriate biochemical indicators and organ function.

Exclusion Criteria:

1. Currently participating in interventional clinical research and treatment, or receiving other research drugs or treatment with research equipment within 4 weeks before the first administration;
2. Accept solid organ or blood system transplantation;
3. Suffer from active autoimmune diseases that require hormone or immunomodulatory treatment, such as rheumatoid arthritis, ankylosing spondylitis, type I diabetes, psoriasis, vitiligo, immune-related thyroid dysfunction, etc. (hormone replacement Can be included after treatment is normal);
4. Suffer from acute or chronic infectious diseases, such as hepatitis B, hepatitis C, tuberculosis, and HIV;
5. Allergic to research drug ingredients;
6. Active infection or fever of unknown cause occurred during the screening period and before the first administration> 38.5℃ (according to the judgment of the investigator, the subject can be included in the group due to fever caused by the tumor);
7. Suffer from uncontrolled clinical symptoms or diseases of the heart, such as:(1) Heart failure above NYHA II; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
8. Suffer from high blood pressure and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
9. Abnormal blood coagulation function (INR>2.0, PT>16s), have a bleeding tendency or are receiving thrombolytic therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin;
10. Obvious coughing up blood or hemoptysis of 10ml or more per day in the 2 months before enrollment;
11. Have significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before enrollment;
12. Have received anti-tumor monoclonal antibodies (mAb) within 4 weeks before using the study drug for the first time, or the adverse events caused by the previously received drug have not recovered (ie ≤ grade 1 or reached the baseline level). Note: Except for subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 hair loss, if the subject has undergone major surgery, the toxic reaction and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
13. The investigator judged other situations not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of radiation pneumonia ≥ grade 2 (1 month, 3 month, 6 month) | up to 6 month
  Incidence rate of radiation pneumonia ≥ grade 2 (1 month, 3 month, 6 month)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 6 month
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
Disease Control Rate （DCR） | up to 6 month
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
6 month progression-free-survival (PFS) rate | up to 6 month
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Treatment-related adverse events | up to 6 month
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No